CLINICAL TRIAL: NCT06805357
Title: Evaluation of Lung Recruitment During Chest Physiotherapy in Mechanically Ventilated Patients
Brief Title: Lung Recruitment During Chest Physiotherapy in Mechanically Ventilated Patients
Acronym: RECRUTKI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: APHP240157
Record Dates: First submitted 2025-01-13; First posted 2025-02-03 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Intensive Care; Invasive Mechanical Ventilation; Chest Physiotherapy; Airway Clearance
Keywords: ICU; Lung recruitment; Respiratory physiotherapy; Rib Cage Compressions (RCC); mechanical ventilation; intensive care

STUDY DESIGN:
Intervention Model Description: The cross-over concerns the ventilatory mode during chest physiotherapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RCC applied in V-ACV (Other): Doest't require description.
  Interventions: Other: Chest Physiotherapy by Rib Cage Compressions (RCC)
- RCC applied in PS (Other): Doest't require description.
  Interventions: Other: Chest Physiotherapy by Rib Cage Compressions (RCC)

INTERVENTIONS:
Other: Chest Physiotherapy by Rib Cage Compressions (RCC) — Bimanual Rib Cage Compressions (RCC) applied to the thorax only, with patients in a standardized position (supine with the head of the bed elevated to 35 degrees). The intervention is standardized in terms of the direction of force (posterior and downward) and the characteristics of the compression (brief and vigorous compressions at the beginning of expiration).

SUMMARY:
In intensive care, respiratory physiotherapy is an integral part of the daily care of patients under invasive mechanical ventilation. Its goals are to improve the clearance of bronchial secretions to allow for the resolution of atelectasis and alveolar recruitment, thereby enhancing respiratory mechanics and gas exchange. The most widespread technique in France is external expiratory compression of the chest.

The effectiveness of this technique depends on the selection of patients (it seems to be more effective in patients with higher secretion levels) and on the practical implementation of the technique (favoring brief and vigorous compressions at the beginning of expiration). However, the effect of the artificial ventilator settings, particularly the ventilatory mode used during the respiratory physiotherapy session, has never been evaluated. The two most commonly used ventilatory modes worldwide are Volume Assist Control Ventilation (V-ACV) and pressure support ventilation (PSV). In this unit, respiratory physiotherapy under artificial ventilation is performed daily on patients with artificial ventilation with abundant secretions, regardless of the ventilatory mode.

DETAILED DESCRIPTION:
It is hypothesized that the effectiveness of respiratory physiotherapy on recruitment depends on the ventilatory mode used during the session.

The primary objective is to compare pulmonary recruitment during respiratory physiotherapy in patients under invasive mechanical ventilation between sessions performed in V-ACV and PSV.

Secondary objectives are to compare the effects of respiratory physiotherapy between V-ACV mode and PSV mode on respiratory mechanics, gas exchange, the amount of drained secretions (weight and volume), the distribution of ventilation, and patient tolerance.

Method:

A cross-over study with a non-invasive physiological endpoint. The primary evaluation criterion is variations in end-expiratory lung volume (ΔEELV) measured 5 minutes before and 5 minutes after a standardized respiratory physiotherapy session in V-ACV or PSV.

The tool used to measure End Expiratory Lung Volume (EELV) is the additional module E-sCOVX of the CARESCAPE R860 ventilator. The procedure is automated and is based on a dilution method.

Secondary outcomes aim to evaluate regional lung ventilation distribution, respiratory mechanics, airway clearance, gas exchange, and patient tolerance.

Tools used to measure secondary evaluation criteria include Electrical Impedance Tomography (EIT) Pulmovista 500® (Dräger), a Pneumotachograph with a pressure transducer inserted in the ventilator circuit (MP150, Biopac Systems, Inc.), and a trap to collect mucus.

The intervention consists of a standardized session in a standardized position (supine at 35° of head elevation).

Each session is composed of 7 series of 3 Rib Cage Compressions (RCC) in a row during each expiration, applied to the thorax only. The interval between the series is about 10 respiratory cycles.

The 2 sessions are done on the same day. One session is performed in the morning, the other in the afternoon. One session is performed in V-ACV and the other in PSV. The order is randomized.

Conclusion:

The results of this study will help better understand the effects of RCC according to the ventilatory mode in patients under invasive mechanical ventilation with mucus excess.

ELIGIBILITY:
Inclusion Criteria:

* Patient under assisted ventilation (in V-ACV or PSV) triggering all ventilator cycles
* Patient deemed " secretive ": requiring ≥ 2 tracheal aspirations every 3 hours
* Patient (or relative) who has given consent to participate in the research
* Patient covered by social security

Exclusion Criteria:

* Age under 18 years
* Legal guardian required
* Recent cardiac and/or thoracic and/or abdominal surgery (< 3 months)
* Rib fracture(s)
* Pneumothorax and/or presence of a chest drain
* Recent neurosurgery (< 3 months) and/or proven or suspected increased intracranial pressure (ICP)
* Hemodynamic instability defined as: noradrenaline ≥ 1mg/h, adrenaline ≥ 0.5 mg/h, dobutamine ≥ 5γ/kg/min.
* Respiratory instability defined as: PEEP > 10 cmH2O and/or PaO2/FiO2 < 150 mm Hg
* Pregnancy
* Hemoptysis
* Sever skin lesions (e.g., burns, Lyell's syndrome)
* Patient under foreign health insurance

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-07-23 (Actual); Primary Completion 2027-06-23 (Estimated); Study Completion 2027-06-23 (Estimated)

PRIMARY OUTCOMES:
Comparison of ΔEELV (after-before) Induced by an RCC Session Performed in V-ACV and PSV | EELV is mesured 5 minutes before, 5 minutes after and 1 hour after each physiotherapy session (morning & afternoon).
  the variation in end-expiratory lung volume (ΔEELV), which refers to the change in the volume of air in the lungs at the end of expiration. This is measured by comparing the end-expiratory lung volume 5 minutes before and 5 minutes after the respiratory physiotherapy session. The ΔEELV is measured in milliliters using the E-sCOVX module of the CARESCAPE R860 ventilator, which employs the nitrogen wash-in/wash-out technique.
Variation in FiO2 During the Session | FiO2 variation is during the physiotherapy session and up to 5 minutes after the session.
  the variation in FiO2 (fraction of inspired oxygen) during the physiotherapy session. FiO2 refers to the percentage of oxygen delivered to the patient through the ventilator. This variation is tracked to assess any changes in the oxygen concentration during the session. The FiO2 variation is expressed as a percentage, with a typical variation of +10% during the procedure, measured using the CARESCAPE R860 ventilator.

SECONDARY OUTCOMES:
Measurement of Airflow in the Ventilator Circuit During Respiratory Physiotherapy Sessions | during and up to 5 minutes after each physiotherapy session
  A pneumotachograph, which measures the flow of air entering and exiting the ventilator circuit, is used for this assessment. The airflow is recorded in liters per minute and provides insight into the volume of air being ventilated during the session. This data is collected using the MP150 Pneumotachograph
mucus volume measurement | measured after each physiotherapy session.
  A mucus collection trap (Cair, LGL) is positioned on the suction line, and the volume of the extracted mucus is precisely measured using a syringe. The volume is recorded in milliliters to assess the amount of mucus cleared during the respiratory physiotherapy session.
Assessment of gas exchange. | 5 minutes before and 5 minutes after each physiotherapy session
  Arterial blood gases are performed only if the patient has an arterial catheter
Assessment of regional lung ventilation distribution. | 5 minutes before, during and 5 minutes after each physiotherapy session.
  Electrical Impedance Tomography (EIT) Pulmovista 500® (Dräger) with the dedicated belt.
Heart rate | 5 minutes before, 5 minutes after and 1 hour after each physiotherapy session.
  quantified in beats per minute (bpm)
Assessment of Airway Pressure Dynamics in the Ventilator Circuit During Respiratory Physiotherapy | during and up to 5 minutes after each physiotherapy session
  A pressure transducer is inserted into the ventilator circuit to measure the airway pressure within the system during the session. This pressure is typically measured in cmH2O. The pressure readings are also analyzed using Acknowledge 5.0 software to evaluate how the airway pressure changes throughout the physiotherapy session.
Quantification of mucus weight | measured after each physiotherapy session.
  the mucus is transferred to a high-precision scale to determine its weight, expressed in grams.
Respiratory rate | 5 minutes before, 5 minutes after and 1 hour after each physiotherapy session.
  expressed in breaths per minute (bpm)
oxygen saturation measurement | 5 minutes before, 5 minutes after and 1 hour after each physiotherapy session.
  measured as a percentage (%)
Blood pressure | 5 minutes before, 5 minutes after and 1 hour after each physiotherapy session.
  Recorded in millimeters of mercury (mmHg)
end-tidal CO2 measurement | 5 minutes before, 5 minutes after and 1 hour after each physiotherapy session.
  measured in millimeters of mercury (mmHg)
Tidal volume | 5 minutes before, 5 minutes after and 1 hour after each physiotherapy session.
  quantified in milliliters (mL), denoting the volume of air inspired or expired during a single respiratory cycle.
minute volume | 5 minutes before, 5 minutes after and 1 hour after each physiotherapy session.
  expressed in liters per minute (L/min), representing the total volume of air ventilating the lungs in one minute.
peak inspiratory pressure | 5 minutes before, 5 minutes after and 1 hour after each physiotherapy session.
  measured in centimeters of water (cmH2O), indicating the maximum pressure reached in the ventilator circuit during the inspiratory phase.
plateau pressure | 5 minutes before, 5 minutes after and 1 hour after each physiotherapy session.
  uantified in centimeters of water (cmH2O), representing the pressure measured at the end of an inspiratory hold, when airflow has ceased.

CONTACTS AND LOCATIONS:
Locations (1):
- Intensive Care Medicine Department Henri Mondor Hospital, Créteil, France

IPD SHARING:
Plan to Share IPD: No
DATAS ARE OWN BY ASSISTANCE PUBLIQUE - HOPITAUX DE PARIS